CLINICAL TRIAL: NCT03408860
Title: Isolating Mechanisms in the Treatment of Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Shannon Sauer Zavala, Research Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3842; K23MH106648-03 (NIH)
Record Dates: First submitted 2018-01-10; First posted 2018-01-24 (Actual); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2-week baseline (Other): Patients complete assessment only for a duration of 2-weeks prior to starting the intervention: Countering Emotional Behaviors Module from the Unified Protocol.
  Interventions: Other: Countering Emotional Behaviors Module from Unified Protocol
- 4-week baseline (Other): Patient complete assessment only for a duration of 4-weeks prior to starting the intervention: Countering Emotional Behaviors Module from the Unified Protocol.
  Interventions: Other: Countering Emotional Behaviors Module from Unified Protocol

INTERVENTIONS:
Other: Countering Emotional Behaviors Module from Unified Protocol — This is a 4-week behavioral treatment that teaches patients to counter problematic emotional avoidance by approaching behaviors and situations that may bring up strong emotions in the short-term, but prevent interfering emotional difficulties in the long-term.

SUMMARY:
Borderline personality disorder (BPD) is a commonly occurring, severe, and costly condition that interferes greatly with quality of life. Considerable comorbidity with other disorders and existing multicomponent treatments with largely untested putative mechanisms of action represent obstacles for effective dissemination of BPD treatment; in light of this gap, the purpose of the present study is to isolate the effects of individual treatment components on putative mechanisms implicated in both BPD. This study will answer important theoretical questions about the mechanism of treatment change, and might lead to more efficacious, cost-effective, and easily disseminable treatment strategies for BPD, a severe and understudied disorder.

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) is a commonly occurring, severe, and costly condition for which treatment efforts have been hindered by several factors. First, extant treatments for BPD are long-term, intensive and consist of multiple components, largely focused on resolving the life-threatening dysregulation that characterizes this disorder. It is important to note, however, that most individuals diagnosed with BPD never attempt suicide or require inpatient hospitalization. Multi-component interventions may not be the most efficient approach for patients with less severe levels of BPD and also make it difficult to draw conclusions regarding which treatment strategies are influencing mechanisms maintaining symptoms. Additionally, extant BPD treatments do no explicitly address high rates of comorbidity with anxiety and depressive disorders; high levels of co-occurrence amongst these disorders underscores the utility of identifying transdiagnostic treatment components relevant to maintaining mechanisms across diagnostic boundaries. The proposed Mentored Patient-Oriented Research Career Development Award (K23) is a four-year plan in support of the applicant's long-term career goal to become a clinical scientist proficient in developing parsimonious, easily disseminated treatments for BPD and other emotional disorders. This project will be completed in two phases. The goal of Phase I, in line with an experimental therapeutics approach, is to investigate the effect of acting inconsistent with emotion-driven behavioral urges on emotional intensity in a sample of individuals diagnosed with BPD in the context of a single-case experiment (alternating treatment design). Phase II will also utilize single-case experimental design (in this case a multiple baseline study) to explore the effects of brief intervention focused solely on acting inconsistent to emotional action tendencies on emotional intensity, tolerance of emotions, and BPD symptoms in a sample diagnosed with BPD. Boston University's Center for Anxiety and Related Disorders, where all research and the bulk of the training activities will take place, is a world-renown clinical research institution with a successful history of treatment development research. Overall, the broader aim of these research and training goals is to address the need for improved treatments for BPD. This study will answer important theoretical questions about the mechanism of treatment change, and might lead to more efficacious, cost-effective, and easily disseminable treatment strategies for BPD, a severe and understudied disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic and Statistical Manual (5th Edition; DSM-5) diagnosis of borderline personality disorder;
2. willing to maintain a stable dose on prescribed psychotropic medication throughout the study duration. This avoids problems with reluctance to discontinue or difficulty with discontinuing, and also the confounding of outcomes from initiation of medication during treatment; this procedure is a longstanding practice at the Center for Anxiety and Related Disorders (CARD) at Boston University for treatment outcome research. Additionally, participants must be
3. fluent in English.

Exclusion Criteria:

In order to maximize generalizability, exclusion criteria are based solely on the well-being of the participant and will consist primarily of conditions that would require prioritization for immediate treatment (e.g., severe suicidality or substance dependence). These include:

1. Current DSM-5 diagnoses of bipolar disorder, schizophrenia, schizoaffective disorder, or organic mental disorder;
2. Clear and current suicidal risk (intent);
3. Current or recent (within 3 months) history of drug dependence;
4. Willingness to refrain from additional psychosocial treatment across the course of the study; and
5. has access to own smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Sauer-Zavala, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University Center for Anxiety and Related Disorders, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2-week Baseline | 4-week Baseline
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2-week Baseline | 4-week Baseline | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Full Range); unit: Years] | 22.67 [19 to 27] | 20.75 [19 to 24] | 21.57 [19 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2 | 3 | 5
  Race: African American | 1 | 0 | 1
  Race: White | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Multidimensional Experiential Avoidance Questionnaire - Distress Aversion Subscale
Description: The Multidimensional Experiential Avoidance Questionnaire - Distress Aversion subscale (MEAQ-DA) assesses aversive reactions to emotional experiences. Total scores representing a sum of items range from 13 to 78, which lower scores indicating more adaptive psychological functioning.
Time Frame: pre-treatment (baseline), post-treatment (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2-week Baseline | 4-week Baseline
Number analyzed (Participants) | 4 | 4
score on a scale
  pre-treatment | 23.21 (7.15) | 23.21 (7.15)
  post-treatment | 19.93 (7.95) | 19.93 (7.95)

2. Secondary Outcome: Zanarini Rating Scale for BPD
Description: The Zanarini Rating Scale for BPD (ZAN-BPD) is a self-report measures that assesses borderline personality disorder symptoms. The total score ranges from 0 to 27 with higher scores representing poorer psychological functioning.
Time Frame: pre-treatment (baseline), post-treatment (4 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2-week Baseline | 4-week Baseline
Number analyzed (Participants) | 4 | 4
score on a scale
  pre-treatment | 9.59 (4.71) | 9.59 (4.71)
  post treatment | 7.12 (5.78) | 7.12 (5.78)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | 2-week Baseline | 4-week Baseline
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT03408860/Prot_SAP_000.pdf